CLINICAL TRIAL: NCT02364427
Title: Arterial Stiffness and Acute Kidney Injury Post-Coronary Artery Bypass Graft Surgery
Brief Title: Arterial Stiffness and AKI Post-CABG
Acronym: Heart-AKI
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KCH heart-AKI
Record Dates: First submitted 2015-02-04; First posted 2015-02-18 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2018-03

CONDITIONS: Acute Kidney Injury
Keywords: Pulse wave velocity; Arterial stiffness; AKI
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arterial stiffness: Arterial stiffness - Vicorder to measure pulse wave velocity
  Interventions: Device: Arterial stiffness - Vicorder to measure pulse wave velocity

INTERVENTIONS:
Device: Arterial stiffness - Vicorder to measure pulse wave velocity — Pulse wave velocity (PWV)measures the stiffness of the arteries. This provides a simple and quick noninvasive method of obtaining the PWV for an arterial segment.
  Other Names: Vicorder

SUMMARY:
Acute Kidney Injury is a condition where your kidneys suddenly stop working properly and usually occurs if you are already unwell with an illness and can happen after having surgery. Having an episode of acute kidney injury increases the risk of progression to chronic kidney disease (CKD) later on and decreases long-term survival. It also has a major socioeconomic impact with regards to admissions and length of hospital stay. There is currently no universally accepted treatment or method of identifying patients that are at risk. The investigators aim to measure arterial stiffness in patients prior to them undergoing cardiac surgery to investigate whether this measurement is associated with an increased risk of patients developing acute kidney injury after surgery. The investigators are planning to measure arterial stiffness, and examine a blood sample, for kidney health-related levels to determine whether there is an association between those patients who have stiff arterial vessels and those patients who may develop acute kidney injury after surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) affects around 20% of all hospitalised patient. Previously it was believed that recovery from an episode of AKI resulted in full renal recovery and return to normal function in the long term. However this assumption may reflect the fact that many of these patients did not receive long term follow-up and a failure to return to their baseline renal function was not identified. It is now recognised that AKI has both major long-term health and socioeconomic impacts. Studies have demonstrated that an episode of AKI can significantly increase both risk of development of chronic kidney disease and early mortality.

Episodes of dialysis-requiring AKI in patients with previously normal renal function who were not dialysis-dependent on discharge resulted in a 28-fold increase in risk of developing severe chronic kidney disease (CKD) stage 4 or 5 and a 2-fold increase in the risk of death at one year when compared to non-AKI controls. This was also observed over a 5-year follow-up period, during which patients who had suffered an episode of AKI were at a 6-fold increased risk of developing both CKD stage 4 or end stage renal failure (ESRF).

There is also an increased risk of death in patients who have experienced an episode of non-dialysis requiring AKI, which remains apparent even with mild AKI stage 1. AKI has a long-term impact on patient morbidity and mortality, an effect that appears to persist despite 'biochemical resolution'. The size of this impact is dependent upon the degree of severity and duration of AKI experienced. However, there is some controversy regarding the link of AKI to CKD. At the present time there is no specific therapy for AKI and the management of patients is completely supportive. Furthermore, in the absence of more sensitive biomarkers, it would appear that even a non-severe episode of AKI already confers a worse prognosis with regards to the risk of development of CKD and long term survival in patients. Thus perhaps focus should be on prevention of AKI as opposed to cure. This is even more pertinent when one considers that the National Confidential Enquiry into Patient Outcomes and Death (NCEPOD) report in 2009 identified 30% of cases as being 'preventable' and a deficiency of care in 50% of cases. The median length of stay for patients diagnosed with AKI was 17.8 days, which was 4.7 days longer than for those without AKI. Marion Kerr, a health economist, reported that by avoiding 'preventable' cases a potential saving of £130-186 million per year could be made.

The difficulty lies in identification of patients that are at risk of AKI. Although factors such as diabetes, older age and low estimated glomerular filtration rate (eGFR) are all associated with increased risk, there is no standardized scoring method for risk. In addition, it is not fully clear why some patients suffer AKI while others, with similar co-morbidities, do not.

Arterial stiffness (AS) is defined as 'the unit of pressure required to generate a change in volume of one unit' within a specified arterial segment. Clinically it can be assessed non-invasively by measurement of pulse wave velocity (PWV. AS varies significantly with age, gender and race, and it is only in the last few years that studies have been undertaken to attempt to quantify a 'normal' or reference value within various populations. Arterial stiffness is also increased in numerous clinical conditions such as diabetes and hypertension and there is now increasing evidence that AS may be an important predictor of disease progression and potential recovery in a wide spectrum of conditions including cardiovascular risk, development of dementia, functional recovery from strokes and in renal disease. Increased AS has been shown to be associated with decreased kidney function and to be an independent risk factor for cardiovascular events in ESRF and in renal transplant recipients.

The mechanism of injury in CKD from increased AS is thought to be related to barotrauma inflicted on glomeruli in a "stiff" vascular system. However, there is little data with regards to the effects of AS in AKI.

For this initial pilot study, we have selected the cohort of patients who are undergoing elective coronary artery bypass graft surgery (CABG) to see if this type of event is associated with increased risk of AKI. On average 450 patients per year undergo CABG surgery at King's College Hospital (KCH) and of these over 200 are elective operations. All elective patients will attend a pre-assessment clinic, which is run weekly with about 20 patients per clinic. Many of these patients will have co-morbidities associated with both an increased risk of AKI and of AS. We have performed a retrospective analysis of incidence of AKI in patients undergoing elective, isolated CABG surgery at KCH from January to December 2012. Of a total of 219 patients, 42 patients were classified as having post-operative AKI according to serum AKI criteria.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing pure (non-valvular repair) CABG surgery
* Male or female
* Aged >18 years
* Written informed consent

Exclusion Criteria:

* Patients who have aortic grafts or renal stents
* Patients at CKD stage 4 or 5 or on dialysis
* Bilateral amputee
* Unable to lie supine for 10-15 mins
* Psychiatric illness, including anxiety, mood and untreated eating disorders
* Infection or course of antibiotics within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing pure (non-valvular repair) CABG surgery
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity (arterial stiffness) | Baseline visit

SECONDARY OUTCOMES:
Kidney function measured by renal blood profile | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sharlene A Greenwood, PhD, Principal Investigator — Consultant renal physiotherapist
Locations (1):
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Greenwood SA, Mangahis E, Castle EM, Wang J, Campbell J, Deshpande R, Jayawardene S. Arterial stiffness is a predictor for acute kidney injury following coronary artery bypass graft surgery. J Cardiothorac Surg. 2019 Mar 7;14(1):51. doi: 10.1186/s13019-019-0873-3. PMID 30845970